CLINICAL TRIAL: NCT03063801
Title: Observational Retrospective Study on the Transfusional Management of the Patients With Congenital Heart Disease Carried Out in Adulthood.
Brief Title: Study on the Transfusional Management of the Patients With Congenital Heart Disease Carried Out in Adulthood.
Status: Completed | Type: Observational
Sponsor: Pierre Wauthy (Other)
Responsible Party: Sponsor-Investigator, Pierre Wauthy, Head of clinic, Brugmann University Hospital
Organization: Brugmann University Hospital (Other)
Other Study IDs: CHUB-transfusion management
Record Dates: First submitted 2017-02-21; First posted 2017-02-24 (Actual); Last update posted 2017-11-22 (Actual); Status verified 2017-11

CONDITIONS: Congenital Heart Defect
Keywords: Congenital Heart Disease; Blood products transfusion
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cardiac surgery: All adult patients having undergone surgery between January 2006 and December 2016 within the CHU Brugmann hospital.
  Interventions: Other: Data extraction in medical files

INTERVENTIONS:
Other: Data extraction in medical files — Data extraction from medical files, countraverified by the bloodbank database for accuracy.

SUMMARY:
Surgeries of heart disease in adulthood can happen in two specific contexts:

* either for an asymptomatic anomaly, possibly coupled with the onset of symptoms later in life and tardily diagnosed and surgically managed
* either for a malformation treated in childhood and requiring a new intervention in adulthood. In recent years, the number of adult patients with congenital heart disease has been steadily increasing. Advances in diagnostic techniques and surgical treatments have enabled many children to reach adulthood. The number of these patients is now higher than the number of children with congenital heart disease. The number of these patients having had surgery in adulthood is also increasing.

Congenital cardiopathies are numerous, ranging from simpler pathologies such as inter-auricular or inter-ventricular communication, to much more complex pathologies such as situations of univentricular hearts. The surgical treatments of these congenital heart diseases are classified into three groups: initial palliative surgery, initial curative surgery or iterative surgery. Palliative surgery aims to improve the clinical tolerance of the patient to the conditions of his pathology or to prevent complications. The curative surgery restores the physiological circulation, the iterative surgery treats a complication or a degeneration appearing after a curative surgery.

Patients undergoing cardiac surgery frequently receive blood products transfusions during the preoperative, intraoperative, or postoperative periods. Several observational studies have shown that in cardiac surgery, the transfusion of blood derivatives is associated with an increase in post-operative morbidity and mortality.

The objective of this study is to analyze the predictive factors of transfusion in congenital patients operated in adulthood at Brugmann University Hospital, depending on the type of surgery applied (palliative, curative or iterative). The secondary objective will be to assess whether there are any differences with the predictive factors identified in non-congenital patients undergoing cardiac surgery, which could potentially alter the transfusion approach in congenital patients.

ELIGIBILITY:
Inclusion Criteria:

Cardiac surgery linked to the presence of a heart congenital malformation.

Exclusion Criteria:

Transfusion refusal from the patient

Min Age: 16 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: All adult patients having had cardiac surgery within the CHU Brugmann hospital, between January 2006 and December 2016.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2017-06-01 (Actual); Study Completion 2017-06-01 (Actual)

PRIMARY OUTCOMES:
Demographic data | 10 years
  Demographic characteristics of the patients (descriptive analysis)
Co-morbidities | 10 years
  List of co-morbidities (descriptive analysis)
Type of surgery | 10 years
  Type of cardiac surgery
Blood loss during surgery | 10 years
  Blood loss during surgery
Complications during surgery | 10 years
  Complications during surgery: descriptive analysis
Complications after surgery | 10 years
  Complications after surgery: descriptive analysis

CONTACTS AND LOCATIONS:
Overall Officials: Aurélie Copin, Principal Investigator — CHU Brugmann; Pierre Wauthy, MD, Study Director — CHU Brugmann
Locations (1):
- CHU Brugmann, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wauthy P, Massaut J, Sanoussi A, Demanet H, Morissens M, Damry N, Dessy H, Malekzadeh-Milani SG, Deuvaert FE. Ten-year experience with surgical treatment of adults with congenital cardiac disease. Cardiol Young. 2011 Feb;21(1):39-45. doi: 10.1017/S1047951110001332. Epub 2010 Oct 6. PMID 20923595
- [Background] Somerville J. Management of adults with congenital heart disease: an increasing problem. Annu Rev Med. 1997;48:283-93. doi: 10.1146/annurev.med.48.1.283. PMID 9046962
- [Background] Society of Thoracic Surgeons Blood Conservation Guideline Task Force; Ferraris VA, Ferraris SP, Saha SP, Hessel EA 2nd, Haan CK, Royston BD, Bridges CR, Higgins RS, Despotis G, Brown JR; Society of Cardiovascular Anesthesiologists Special Task Force on Blood Transfusion; Spiess BD, Shore-Lesserson L, Stafford-Smith M, Mazer CD, Bennett-Guerrero E, Hill SE, Body S. Perioperative blood transfusion and blood conservation in cardiac surgery: the Society of Thoracic Surgeons and The Society of Cardiovascular Anesthesiologists clinical practice guideline. Ann Thorac Surg. 2007 May;83(5 Suppl):S27-86. doi: 10.1016/j.athoracsur.2007.02.099. PMID 17462454
- [Background] Wilkinson KL, Brunskill SJ, Doree C, Trivella M, Gill R, Murphy MF. Red cell transfusion management for patients undergoing cardiac surgery for congenital heart disease. Cochrane Database Syst Rev. 2014 Feb 7;2014(2):CD009752. doi: 10.1002/14651858.CD009752.pub2. PMID 24510598
- [Background] Mulaj M, Faraoni D, Willems A, Sanchez Torres C, Van der Linden P. Predictive factors for red blood cell transfusion in children undergoing noncomplex cardiac surgery. Ann Thorac Surg. 2014 Aug;98(2):662-7. doi: 10.1016/j.athoracsur.2014.04.089. Epub 2014 Jun 24. PMID 24968768
- [Background] Zomer AC, Verheugt CL, Vaartjes I, Uiterwaal CS, Langemeijer MM, Koolbergen DR, Hazekamp MG, van Melle JP, Konings TC, Bellersen L, Grobbee DE, Mulder BJ. Surgery in adults with congenital heart disease. Circulation. 2011 Nov 15;124(20):2195-201. doi: 10.1161/CIRCULATIONAHA.111.027763. Epub 2011 Oct 10. PMID 21986279
- [Background] Loup O, von Weissenfluh C, Gahl B, Schwerzmann M, Carrel T, Kadner A. Quality of life of grown-up congenital heart disease patients after congenital cardiac surgery. Eur J Cardiothorac Surg. 2009 Jul;36(1):105-11; discussion 111. doi: 10.1016/j.ejcts.2009.03.023. Epub 2009 May 12. PMID 19442530